CLINICAL TRIAL: NCT05323084
Title: A Cross-over Pilot Trial to Determine the Effect of an LSU Patented Dietary Herbal Supplement on Quality of Life
Brief Title: Effect of a Dietary Supplement on Quality of Life
Acronym: SleepLift
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Principal Investigator, Frank Greenway, Professor, Chief Medical Officer, Pennington Biomedical Research Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: PBRC 2020-039
Record Dates: First submitted 2022-03-27; First posted 2022-04-12 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-11

CONDITIONS: Quality of Life
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Intervention Model Description: 1 week of treatment with a three component supplement or a placebo in people with insomina on two occasions separated by a 2-week washout
Who Masked: Participant, Care Provider, Investigator
Masking Description: Liquid that looks and tastes the same, but only one has the three food components. The order in which the subjects get the 3-component supplement and the placebo is randomly assigned and balanced.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary supplement (Experimental): Green tea extract 5 grams, Chicory extract 1gram and collagen peptides 5 grams in 60ml with sugar, erythritol and 2% potassium sorbate and 1% flavor
  Interventions: Dietary Supplement: Dietary supplement
- Placebo (Placebo Comparator): 60ml of water, sugar, erythritol, 2% potassium sorbate, and 1% flavor
  Interventions: Dietary Supplement: Dietary supplement

INTERVENTIONS:
Dietary Supplement: Dietary supplement — 1 week of each intervention at bedtime with a 2-week washout period in between interventions
  Other Names: Placebo

SUMMARY:
The purpose of this research study is to evaluate the effect of a combination of 3 food components to improve the quality of life in people who have trouble sleeping. Ten subjects with insomnia will drink 2 ounces of the supplement or a placebo for 1 week and after a 2 weeks washout period, will take the treatment they did not take the first week. Questionnaires to evaluate quality of life, and a sleep study will be done before and after each treatment week.

DETAILED DESCRIPTION:
Each participant will be in the study for about 1 month. The questionnaires consist of Chubon Quality of Life Rating, the Multi-dimensional Fatigue Inventory, Insomnia Severity Index, the Epworth Sleepiness, Pittsburgh Sleep Quality Index. Subjects will be screened with a medical questionnaire, vital signs, height, weight, oximetry to identify sleep apnea, a CBC and chemistry panel and the Insomnia severity Index. Weight, vital signs, adverse event questioning, dispensing and collection of test material will be done at each visit. During each treatment week subjects will wear an actigraph, keep a sleep diary and at the beginning and end of each treatment week subjects will have a polysomnography. At the end of each treatment period subjects will have a chemistry panel, a CBC, and a buffy coat will be archived.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or women >50 years of age
* Usual bedtime between 9pm and midnight
* Insomnia for >6months by ICSD-2 criteria
* Insomnia Severity Index score >10 and Sleep-onset latency or Waking after sleep onset >30 minutes

Exclusion Criteria:

* Have diabetes mellitus
* Taking chronic medication not on a stable dose for >1month
* Taking sedating or hypnotic medications
* Have a sleep disorder other than insomnia (like sleep apnea) Adults unable to consent Prisoners Pregnant women Individuals not yet adults

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-02-25 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2022-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula R Brantley, PhD, Study Chair — Pennington Biomedical Research Center Institutional Review Board
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available on approval of the PI
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Study is expected to be done and report generated by June 2022
Access Criteria: Data can be accessed, if the use is approved by the PI

REFERENCES:
- See also: Chubon Quality of Life Rating, — https://pubmed.ncbi.nlm.nih.gov/11438246/
- See also: Validation of the Insomnia Severity Index — https://pubmed.ncbi.nlm.nih.gov/11438246/
- See also: Epworth Sleepiness scale — https://pubmed.ncbi.nlm.nih.gov/1798888/
- See also: Pittsburgh Sleep Quality Index — https://pubmed.ncbi.nlm.nih.gov/2748771/

RESULTS

PARTICIPANT FLOW:
Groups:
- Dietary Supplement First and Placebo Second: Green tea extract 5 grams, Chicory extract 1gram and collagen peptides 5 grams in 60ml with sugar, erythritol and 2% potassium sorbate and 1% flavor
  Dietary supplement: 1 week of each intervention at bedtime with a 2-week washout period in between interventions
- Placebo First Dietary Supplement Second: 60ml of water, sugar, erythritol, 2% potassium sorbate, and 1% flavor
  Dietary supplement: 1 week of each intervention at bedtime with a 2-week washout period in between interventions
Period: Period 1
Arm/Group | Dietary Supplement First and Placebo Second | Placebo First Dietary Supplement Second
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Period 2 - Washout
Arm/Group | Dietary Supplement First and Placebo Second | Placebo First Dietary Supplement Second
Started | 5 | 5 (One participant was lost to follow-up during the wash-out period.)
Completed | 5 | 4
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: Period 3
Arm/Group | Dietary Supplement First and Placebo Second | Placebo First Dietary Supplement Second
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Baseline Characteristic of Study Participant: Characteristics of the study participant prior to any intervention
Arm/Group | Baseline Characteristic of Study Participant
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Body mass index [Mean (Standard Deviation); unit: kg per meter square] | 30 (10)
Glucose [Mean (Standard Deviation); unit: mg/dL] | 98 (14)
Wake after sleep onset [Mean (Standard Deviation); unit: minutes] — Wake after sleep onset is determined by 7-day accelerometry and measures total number of minutes a person is awake after having initially fallen asleep in min. Higher values indicate poor sleep.
  minutes | 75 (33)
Insomnia severtiy index [Mean (Standard Deviation); unit: scores on a scale.] — Insomnia severity index ranges from 0 to 28. Scores above 15 are considered to be clinically significant insomnia.
  scores on a scale. | 21 (4)

OUTCOME MEASURES:

1. Primary Outcome: Chubon Lifestyle Score
Description: Total score ranges from 20 to 140 with higher scores being better quality of life
Time Frame: 1 week
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Dietary Supplement | Placebo
Number analyzed (Participants) | 9 | 10
score on a scale
  Baseline | 103.9 (2.5) | 100.9 (2.4)
  Follow up | 100.4 (2.5) | 102.9 (2.4)

2. Secondary Outcome: Pittsburgh Sleep Quality Index Score
Description: Total Score ranges from 0 to 21 with higher sleep quality having lower numerical values
Time Frame: 1 week
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Dietary Supplement | Placebo
Number analyzed (Participants) | 9 | 10
score on a scale
  Baseline | 10.8 (1) | 10.5 (1.0)
  Follow-up | 9.1 (1) | 8.3 (1)

3. Secondary Outcome: Epworth Sleepiness Scale
Description: Total Score score 0-24 with higher scores having greater degree of sleepiness
Time Frame: 1 week
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Dietary Supplement | Placebo
Number analyzed (Participants) | 9 | 10
score on a scale
  Baseline | 8.4 (1.2) | 8.8 (1.2)
  Follow up | 9.9 (1.2) | 6.9 (1.2)

4. Secondary Outcome: Multidimensional Fatigue Index -General Fatigue
Description: Index of self-perceived general fatigue. Score range from 4 to 20 with high score indicative of more fatigue.
Time Frame: 1-week
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Dietary Supplement | Placebo
Number analyzed (Participants) | 9 | 10
score on a scale
  Baseline | 15.1 (1.0) | 14.7 (1.0)
  Follow-up | 14.0 (1.0) | 13.4 (1.0)

5. Secondary Outcome: Multidimensional Fatigue Index - Physical Fatigue
Description: Index of self-perceived physical fatigue. Score range of 4 to 20 with higher score indicative more fatigue.
Time Frame: 1 week
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Dietary Supplement | Placebo
Number analyzed (Participants) | 9 | 10
score on a scale
  Baseline | 11.1 (1.3) | 10.3 (1.3)
  Follow up | 9.5 (1.3) | 11.3 (1.3)

6. Secondary Outcome: Multidimensional Fatigue Index - Mental Fatigue
Description: Index of self-perceived mental fatigue. Score ranges from 4 to 20 with higher scores indicative of more fatigue.
Time Frame: 1 week
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Dietary Supplement | Placebo
Number analyzed (Participants) | 9 | 10
score on a scale
  Baseline | 11.7 (1) | 12.5 (1)
  Follow-up | 12.4 (1) | 11.7 (1)

7. Other Pre Specified Outcome: Sleep Latency
Description: Determined by Polysomnography - time it takes for a person to fall asleep in min
Time Frame: 1-week
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Dietary Supplement | Placebo
Number analyzed (Participants) | 9 | 10
Minutes
  Baseline | 28 (8) | 32 (8)
  Follow-up | 24 (8) | 28 (8)

8. Other Pre Specified Outcome: Wake After Sleep Onset
Description: Determined by polysomnography - total number of minutes a person is awake after having initially fallen asleep in min.
Time Frame: 1-week
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Dietary Supplement | Placebo
Number analyzed (Participants) | 9 | 10
Minutes
  Baseline | 77 (21) | 71 (20)
  Follow-up | 79 (21) | 72 (20)

9. Other Pre Specified Outcome: Sleep Efficiency
Description: Determined by polysomnography - ratio of the total time spent asleep in a night compared to the total time spent in bed in percentage.
Time Frame: 1-week
Measure: Least Squares Mean (Standard Error); unit: % of total sleep time
Arm/Group | Dietary Supplement | Placebo
Number analyzed (Participants) | 9 | 10
% of total sleep time
  Baseline | 80 (4) | 80 (4)
  Follow-up | 80 (4) | 81 (4)

ADVERSE EVENTS:
Time Frame: up to 8 weeks
Arm/Group | Dietary Supplement | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 0/9 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-23): https://cdn.clinicaltrials.gov/large-docs/84/NCT05323084/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-23): https://cdn.clinicaltrials.gov/large-docs/84/NCT05323084/ICF_001.pdf